CLINICAL TRIAL: NCT04944745
Title: Myofascial Release of the Pectoral Fascia: Effect on Shoulder Posture, Muscle Length, Muscle Activity, and Movement Performance
Brief Title: Myofascial Release of the Pectoral Fascia
Acronym: MTRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Centennial College (Other)
Responsible Party: Principal Investigator, Trisha Scribbans, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 50187
Record Dates: First submitted 2021-06-02; First posted 2021-06-30 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Single blind between subjects repeated measures crossover design
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants will have knowledge of the two different intensity treatments they will receive. However, the researchers will be blinded as to which treatment intensity the participant received at which session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release (MFR) (Experimental): The pectoral MFR will be completed by an experienced registered massage therapist (RMT). They will stand on the participant's right side slightly rotated to the left facing towards the participant's left hip and apply a cross-hand MFR technique to the superficial pectoral fascia on the right side. The therapist will begin by placing the distal region of the anterior palm of the anchoring hand (therapist's right hand) on the right edge of the anterior sternum at the level of the 3rd to the 6th ribs on the skin and the draping over the pectoral fascia. They will then apply a gentle posterior pressure to hold the fascia in place. The forearm of the mobilizing hand (RMT's left hand) will be directed to the right shoulder wit hate right forearm crossing over the left and the contact of are of the mobilizing hand will be the skin superficial to the pectoral fascia and insertion of pectorals major on the anterior aspect of the humerus. This will be held for four minutes.
  Interventions: Other: Myofascial Release
- Soft-touch Control (CON) (Sham Comparator): This control treatment will be set up the same way in regards to the RMT's hand placement, except no pressure will be applied. The RMT's hands will simply be resting over the contact points. This treatment will also be held for four minutes.
  Interventions: Other: Soft-touch Control

INTERVENTIONS:
Other: Myofascial Release — Moderate pressure manual treatment to the pectoral fascia.
  Arms: Myofascial release (MFR)
Other: Soft-touch Control — No pressure manual treatment to the pectoral fascia.
  Arms: Soft-touch Control (CON)

SUMMARY:
Neck-shoulder pain is among the most common health care problems, especially in office workers and females. Forward shoulder posture (FSP) is a common postural deviation and known risk factor for the development of neck-shoulder pain and pathology. Common approaches for reducing FSP include stretching and performing manual techniques to increase the length and extensibility of the scapular protractors, and strengthening the scapular retractors. Myofascial release (MFR) is a group of manual techniques that elongate and soften restricted fascia, however, the effects of myofascial release to the pectorals on FSP are currently unknown. The objectives of this study are to determine the impact of 4-minutes of MFR on: 1) FSP, 2) pectoral length, 3) muscle activity of the upper, middle, and lower trapezius and pectoralis major, 4) scapular retractor to protractor ratio of activity, and 4) movement performance compared to a soft-touch control. We hypothesize that MFR will: 1) decrease FSP, 2) increase pectoral length, 3) increase upper, middle, and lower trapezius activity and decrease pectorals major activity, 4) increase the scapular retractor to protractor ratio of activity, and 4) improve movement performance.

ELIGIBILITY:
Inclusion Criteria:

* have 1 cm of anterior deviation of the acromion process (forward shoulder posture)
* right handed

Exclusion Criteria:

* recent history (<6 months) of neck, shoulder, or upper back pain
* recent history (<6 months) of neck, shoulder, or upper back injury/pathology
* history of orthopaedic or neurological disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Change in Forward shoulder posture after intervention | 30-minutes
  Relative- photographic analysis. Participant stand in a relaxed position and have a photo taken from their side where an online program will be used to quantify their forward shoulder posture
Change in Forward shoulder posture after intervention | 30-minutes
  Absolute measurements taken- double square method. Participants will stand with their back against the wall and the tool will measure the distance from the wall to their acromion process.
Change in Pectoral Length after intervention | 30-minutes
  Measured passive horizontal abduction of the shoulder
Change in Muscle Activity- Upper Trapezius after intervention | 30-minutes
  sEMG during a reaching task
Change in Muscle Activity- Middle Trapezius after intervention | 30-minutes
  sEMG during a reaching task
Change in Muscle Activity- Lower Trapezius after intervention | 30-minutes
  sEMG during a reaching task
Change in Muscle Activity- Pectoralis Major after intervention | 30-minutes
  sEMG during a reaching task
Change in Movement performance- reaction time after intervention | 30-minutes
  Participants will complete a reaching task using custom designed software (E-Prime). The reaching task is a modified Fitts' Task where the participant must reach towards one of five randomly appearing targets.
Change in Movement performance- movement time after intervention | 30-minutes
  Participants will complete a reaching task using custom designed software (E-Prime). The reaching task is a modified Fitts' Task where the participant must reach towards one of five randomly appearing targets.
Change in Movement performance- accuracy after intervention | 30-minutes
  Participants will complete a reaching task using custom designed software (E-Prime). The reaching task is a modified Fitts' Task where the participant must reach towards one of five randomly appearing targets.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chimera NJ, Bohunicky S, Glazebrook C, Scribbans T. Postural factors contributing to reaching speed and accuracy. Int J Occup Saf Ergon. 2025 Sep;31(3):903-912. doi: 10.1080/10803548.2025.2466919. Epub 2025 Mar 10. PMID 40062388